CLINICAL TRIAL: NCT03259009
Title: Predictive Impact of RAS Mutations in Circulating Tumor DNA for Efficacy of Anti-EGFR Reintroduction Treatment in Patients With Metastatic Colorectal Cancer
Brief Title: RAS Mutations in ctDNA and Anti-EGFR reINTROduction in mCRC (RASINTRO)
Acronym: RASINTRO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Association des Gastroentérologues Oncologues (Other)
Collaborators: Hôpital Européen George Pompidou, APHP, Paris, France (Unknown); UMR-S1147, Université Paris Descartes (Unknown); Methodology and Quality of Life in Oncology Unit, Besançon University Hospital, France (Unknown); Pitié-Salpêtrière Hospital (Other); Poitiers University Hospital, Poitiers, France (Unknown); University Hospital Robert Debré, Reims, France (Unknown); Rennes University Hospital, Rennes, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RASINTRO
Record Dates: First submitted 2017-08-14; First posted 2017-08-23 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; anti-EGFR therapy; rechallenge; circulating tumor DNA; biomarker; RAS mutations
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Circulating tumor DNA
  During the inclusion period, a blood sample will be taken just before the first 3 cycles of chemotherapy (C1, C2 and C3) and at tumor progression for mCRC patients treated in one of the participating AGEO centers. These samples will not require any additional invasive procedures since they will be made from the Huber needle previously implanted in the catheter for previously scheduled chemotherapy cycles.
  The patient will sign an information letter and a specific informed consent for blood collection and biological studies. In case of specific refusal, the patient will not be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with metastatic colorectal cancer: Rechallenge with an anti-EGFR monoclonal antibody in patients with metastatic colorectal cancer

SUMMARY:
Some data have suggested a clinical survival benefit related to the reintroduction of anti-EGFRs therapy in patients with metastatic colorectal cancer (mCRC). Based on resistance mechanisms related to the development of resistant clones, the investigators could assume that patients who benefited most from the reintroduction of anti-EGFRs were those who, through interval chemotherapy, had no longer mutated RAS clone in plasma that appeared during the progression with the first anti-EGFR treatment. Conversely, those who did not benefit from this therapy were probably patients who had mutated RAS clones circulating at the time of reintroduction of anti-EGFRs. To support this hypothesis, investigators propose to evaluate the correlation between the eventual presence of RAS mutations in circulating blood and the efficacy of an anti-EGFR therapy reintroduction in patients with mCRC.

DETAILED DESCRIPTION:
Somatic mutations in KRAS exon 2 are considered as a predictive marker of lack of efficacy for anti-EGFR therapy (panitumumab or cetuximab) in patients with metastatic colorectal cancer. Recently, it has been shown that rare mutations of KRAS (exons 3 or 4) or NRAS (exons 2, 3 and 4) were also predictive for resistance to anti-EGFR antibodies. These data led to a further restriction of anti-EGFR therapy to the subgroup of patients without any RAS mutations.

Emerging RAS mutations in circulating tumor DNA (ctDNA) could be detected in patients with RAS non-mutated colorectal cancer treated with anti-EGFR. The appearance in blood of these rare RAS mutated clones during anti-EGFR therapy was associated with shorter progression free-survival. These results suggest that the growing and development of rare RAS mutated clone, which is probably pre-existing in the primary tumor, may constitute a mechanism of resistance for anti-EGFR therapy.

A phase II prospective study has evaluated the interest of reintroduction of cetuximab in 39 patients previously treated with irinotecan and cetuximab. For inclusion, patients should have had a clinical benefit (stable disease for at least 6 months or clinical response) with the previous line of cetuximab plus irinotecan therapy and then a progression disease for which underwent a new line of chemotherapy before the rechallenge of cetuximab plus irinotecan. The median number of line of chemotherapy before inclusion was 4, and the median interval time between last cycle of first cetuximab-based therapy and first cycle of the retreatment was 6 months. In this study, the overall response rate was 53.8%, and the median progression free-survival was 6.6 months. No evaluation of circulating tumor DNA was performed in this study.

These data indicate that the colorectal cancer genome adapts dynamically to intermittent drug schedules and provide a molecular explanation for the efficacy of rechallenge therapies based on EGFR blockage. It seems that efficacy of anti-EGFR reintroduction could be specifically observed in subgroup of patients who no longer have a RAS mutated clone following the interval chemotherapy.

The aim of this prospective non-interventional study is to evaluate the predictive impact of RAS mutations in circulating tumor DNA for efficacy of anti-EGFR reINTROduction (RASINTRO study) treatment in patients with metastatic colorectal cancer.

The primary endpoint will be the correlation between RAS mutations status in circulating tumor DNA and progression-free survival from the reintroduction of anti-EGFR therapy.

The blood sample for circulating tumor DNA assessment will be carried out in patients who agreed to participate in this observational study just before the first 3 cycles of chemotherapy. This study does not require any additional invasive procedures to those already scheduled for routine care. Indeed, blood sample will be collected from the Huber needle previously implanted in the port-a-cath for chemotherapy perfusion.

After DNA extraction from bood samples, RAS mutation testing will be performed using sequencing with a panel of genes (Ion AmpliSeq Colon and Lung Cancer Panel).

The data related to the patient (age at diagnosis, sex, weight, height, WHO performance status), tumor (tumor markers CEA and CA 19-9, histological type and tumor differentiation, tumor stage, and metastatic sites) and treatment (resection of the primary tumor, date of surgery, lines of chemotherapy, protocol regimen) will be collected anonymously. Monitoring data concern the efficacy of chemotherapy (tumor response, the date of disease progression/death).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Metastatic colorectal cancer histological confirmed without somatic mutations of KRAS (exons 2, 3 et 4) and NRAS (exons 2, 3 et 4)
* Apart from contraindication, patients should have already received fluoropyrimidine, irinotecan, oxaliplatin, anti-EGFR (panitumumab or cetuximab) and anti-angiogenic (bevacizumab or aflibercept) therapies
* Previous treatment with anti-EGFR-based chemotherapy (panitumumab or cetuximab) should have provided an objective tumor response (according to RECIST 1.1 criteria) and/or PFS ≥ 4 months.
* At least one line of interval chemotherapy between the last cycle of anti-EGFR based treatment and reintroduction of anti-EGFR therapy
* Signed written informed consent obtained prior to any study specific screening procedures

Exclusion Criteria:

* Discontinuation of first anti-EGFR therapy for other reasons than tumor progression
* Previous malignancy other than colorectal cancer in the last 5 years
* Medical, sociological, psychological or legal conditions that would not permit the patient to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer receiving a reintroduction of anti-EGFR monoclonal antibody alone (without any associated antitumor drugs)
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from the date of beginning the reintroduction of anti-EGFR therapy to date of tumor progression or death from any cause, whichever occurred first, assessed up to 6 months.
  PFS will be evaluated according to the RAS mutations on circulating tumor DNA status

SECONDARY OUTCOMES:
Tumor response | The tumor response will be assessed in patients with measurable lesions according to RECIST criteria version 1.1, assessed up to 6 months
  Tumor response will be evaluated according to the RAS mutations on circulating tumor DNA
Overall survival (OS) | Time from the date of beginning the reintroduction of anti- EGFR therapy to date of death of any cause, through study completion, an average of 1 year
  OS will be evaluated according to the RAS mutations on circulating tumor DNA

CONTACTS AND LOCATIONS:
Overall Officials: Aziz ZAANAN, MD, PhD, Principal Investigator — European Georges Pompidou Hospital, Paris, France; Julien TAIEB, MD, PhD, Study Chair — European Georges Pompidou Hospital, Paris, France; Pierre LAURENT-PUIG, MD, PhD, Study Director — UMR-S1147, Université Paris Descartes, Paris, France

REFERENCES:
- [Result] Van Cutsem E, Kohne CH, Hitre E, Zaluski J, Chang Chien CR, Makhson A, D'Haens G, Pinter T, Lim R, Bodoky G, Roh JK, Folprecht G, Ruff P, Stroh C, Tejpar S, Schlichting M, Nippgen J, Rougier P. Cetuximab and chemotherapy as initial treatment for metastatic colorectal cancer. N Engl J Med. 2009 Apr 2;360(14):1408-17. doi: 10.1056/NEJMoa0805019. PMID 19339720
- [Result] Douillard JY, Siena S, Cassidy J, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Oliner KS, Wolf M, Gansert J. Randomized, phase III trial of panitumumab with infusional fluorouracil, leucovorin, and oxaliplatin (FOLFOX4) versus FOLFOX4 alone as first-line treatment in patients with previously untreated metastatic colorectal cancer: the PRIME study. J Clin Oncol. 2010 Nov 1;28(31):4697-705. doi: 10.1200/JCO.2009.27.4860. Epub 2010 Oct 4. PMID 20921465
- [Result] Amado RG, Wolf M, Peeters M, Van Cutsem E, Siena S, Freeman DJ, Juan T, Sikorski R, Suggs S, Radinsky R, Patterson SD, Chang DD. Wild-type KRAS is required for panitumumab efficacy in patients with metastatic colorectal cancer. J Clin Oncol. 2008 Apr 1;26(10):1626-34. doi: 10.1200/JCO.2007.14.7116. Epub 2008 Mar 3. PMID 18316791
- [Result] Karapetis CS, Khambata-Ford S, Jonker DJ, O'Callaghan CJ, Tu D, Tebbutt NC, Simes RJ, Chalchal H, Shapiro JD, Robitaille S, Price TJ, Shepherd L, Au HJ, Langer C, Moore MJ, Zalcberg JR. K-ras mutations and benefit from cetuximab in advanced colorectal cancer. N Engl J Med. 2008 Oct 23;359(17):1757-65. doi: 10.1056/NEJMoa0804385. PMID 18946061
- [Result] Douillard JY, Oliner KS, Siena S, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Williams R, Rong A, Wiezorek J, Sidhu R, Patterson SD. Panitumumab-FOLFOX4 treatment and RAS mutations in colorectal cancer. N Engl J Med. 2013 Sep 12;369(11):1023-34. doi: 10.1056/NEJMoa1305275. PMID 24024839
- [Result] Van Cutsem E, Lenz HJ, Kohne CH, Heinemann V, Tejpar S, Melezinek I, Beier F, Stroh C, Rougier P, van Krieken JH, Ciardiello F. Fluorouracil, leucovorin, and irinotecan plus cetuximab treatment and RAS mutations in colorectal cancer. J Clin Oncol. 2015 Mar 1;33(7):692-700. doi: 10.1200/JCO.2014.59.4812. Epub 2015 Jan 20. PMID 25605843
- [Result] Misale S, Yaeger R, Hobor S, Scala E, Janakiraman M, Liska D, Valtorta E, Schiavo R, Buscarino M, Siravegna G, Bencardino K, Cercek A, Chen CT, Veronese S, Zanon C, Sartore-Bianchi A, Gambacorta M, Gallicchio M, Vakiani E, Boscaro V, Medico E, Weiser M, Siena S, Di Nicolantonio F, Solit D, Bardelli A. Emergence of KRAS mutations and acquired resistance to anti-EGFR therapy in colorectal cancer. Nature. 2012 Jun 28;486(7404):532-6. doi: 10.1038/nature11156. PMID 22722830
- [Result] Morelli MP, Overman MJ, Dasari A, Kazmi SMA, Mazard T, Vilar E, Morris VK, Lee MS, Herron D, Eng C, Morris J, Kee BK, Janku F, Deaton FL, Garrett C, Maru D, Diehl F, Angenendt P, Kopetz S. Characterizing the patterns of clonal selection in circulating tumor DNA from patients with colorectal cancer refractory to anti-EGFR treatment. Ann Oncol. 2015 Apr;26(4):731-736. doi: 10.1093/annonc/mdv005. Epub 2015 Jan 26. PMID 25628445
- [Result] Siravegna G, Mussolin B, Buscarino M, Corti G, Cassingena A, Crisafulli G, Ponzetti A, Cremolini C, Amatu A, Lauricella C, Lamba S, Hobor S, Avallone A, Valtorta E, Rospo G, Medico E, Motta V, Antoniotti C, Tatangelo F, Bellosillo B, Veronese S, Budillon A, Montagut C, Racca P, Marsoni S, Falcone A, Corcoran RB, Di Nicolantonio F, Loupakis F, Siena S, Sartore-Bianchi A, Bardelli A. Clonal evolution and resistance to EGFR blockade in the blood of colorectal cancer patients. Nat Med. 2015 Jul;21(7):795-801. doi: 10.1038/nm.3870. Epub 2015 Jun 1. PMID 26030179
- [Result] Santini D, Vincenzi B, Addeo R, Garufi C, Masi G, Scartozzi M, Mancuso A, Frezza AM, Venditti O, Imperatori M, Schiavon G, Bronte G, Cicero G, Recine F, Maiello E, Cascinu S, Russo A, Falcone A, Tonini G. Cetuximab rechallenge in metastatic colorectal cancer patients: how to come away from acquired resistance? Ann Oncol. 2012 Sep;23(9):2313-2318. doi: 10.1093/annonc/mdr623. Epub 2012 Mar 5. PMID 22396447
- [Result] Norton SE, Lechner JM, Williams T, Fernando MR. A stabilizing reagent prevents cell-free DNA contamination by cellular DNA in plasma during blood sample storage and shipping as determined by digital PCR. Clin Biochem. 2013 Oct;46(15):1561-5. doi: 10.1016/j.clinbiochem.2013.06.002. Epub 2013 Jun 13. PMID 23769817
- [Derived] Zaanan A, Bergen ES, Evesque L, Meurisse A, Artru P, Lecomte T, Bouche O, Lepere C, Ambrosini M, Coriat R, Lievre A, Cohen R, Boige V, Louafi S, Bachet JB, Goyer S, Taieb J, Vernerey D, Blons H, Laurent-Puig P. Circulating tumor DNA driving anti-EGFR rechallenge therapy in metastatic colorectal cancer: the RASINTRO prospective multicenter study. J Natl Cancer Inst. 2025 Nov 1;117(11):2362-2371. doi: 10.1093/jnci/djaf229. PMID 40833930